CLINICAL TRIAL: NCT00940914
Title: Evaluation of Radioligand Uptake (FP-CIT) of Dopamine Transporters in Patients Suffering From Parkinson's Disease With or Without Pain
Brief Title: Dopaminergic Loss and Pain in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0730302; AOL 2007
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease; Pain
Keywords: Parkinson's disease; pain; dopamine transporters imaging
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — ioflupane; 2-carbomethoxy-8-(3-fluoropropyl)-3-(4-iodophenyl)tropane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pain disorders (Other): patients with Parkinson's disease presenting pain disorders
  Interventions: Drug: ioflupane 123I (DATSCAN®)
- without pain disorders (Other): patients with Parkinson's disease without pain disorders
  Interventions: Drug: ioflupane 123I (DATSCAN®)

INTERVENTIONS:
Drug: ioflupane 123I (DATSCAN®) — One administration (2,5 ml) of ioflupane 123I 0,07-0,13 µg/ml; 74 MBq/ml; IV (in the vein)
  Other Names: - N-w-fluoropropyl-2beta-carbomethoxy-3beta-(4-iodophenyl)tropane; - FP-CIT

SUMMARY:
About 46% of patients suffering from Parkinson's disease present pain disorders. Parkinson disease is characterized by loss of dopaminergic neurons. The aim of this study is to assess the relationship between the loss of dopaminergic neurons and the existence of pain in Parkinson's disease. Using single photon emission computerized tomography (SPECT) imaging (123I FP-CIT, which binds dopamine transporter) and the determination of subjective pain threshold, the investigators will establish correlations between dopaminergic degeneration and pain perception.

DETAILED DESCRIPTION:
Parkinson's disease is a frequent neurodegenerative disease leading to motor handicap, cognitive and pain disorders. These pain disorders could be correlated to dopaminergic loss.

The clinical trial will be conducted in a single center (Neurology Department, Purpan Hospital, Toulouse, France). The study is classified as a physiopathology one. Twenty patients with Parkinson's disease, presenting pain disorders or not, will be selected. This clinical trial will last one year. All the exams, including image acquisition will be done the same day. These will take about 6 hours for each patient.

Expected results: Binding of 123I FP-CIT to dopamine transporters should negatively correlate with pain intensity and also with thermal pain thresholds in patients suffering from Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically established Parkinson's disease according to the UKPDSBB (UK Parkinson's Disease Society Brain Bank) (Gibb et Less, 1998; Hugues et al, 1992).
* Male or Female patients, aged from 30 to 70 years.
* Patients must benefit from the French Social security system.
* Patients must give a written informed consent.
* Female fertile patients must use an efficient method of contraception.

If patients suffer from chronic pain, pain must be related to Parkinson's disease.

Exclusion Criteria:

* Patients with a syndrome other than the idiopathic Parkinson's disease.
* Patients suffering from important trembling during the OFF periods or abnormal involuntary movements (dyskinesia) during the ON periods, not allowing the imagery exam to be performed.
* Patients suffering from another disease causing chronic pain.
* Patients suffering from cancer.
* Patients with cognitive dysfunction.
* Patients not able to complete the scales.
* Pregnant, breastfeeding or fertile female patients not using an efficient method of contraception.
* Patients not willing to participle in the trial.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Single photon emission computerized tomography (SPECT) will be used to evaluate binding of 123I FP-CIT to dopamine transporters. This exam will allow calculation of the ratio of specific to non specific binding of 123I FP-CIT to dopamine transporters. | Image acquisition (SPECT) will be performed after three hours post-injection of 123I FP-CIT.
Pain perception will be evaluated by the determination of subjective pain thresholds (thermal pain thresholds, thermotest). A thermode will be used to determine the heat and cold pain thresholds. | Image acquisition (SPECT) will be performed after three hours post-injection of 123I FP-CIT.

SECONDARY OUTCOMES:
Severity of Parkinson's disease will be evaluated with the Unified Parkinson's disease Rating Scale (UPDRS) and the Hoehn and Yahr scale | Evaluation will be done within three hours before image acquisition (SPECT).
Short French version of McGill pain questionnaire (MPQ). | Evaluation will be done within three hours before image acquisition (SPECT).
Pain intensity will be assessed using a 10 cm visual analogue scale (VAS) (0 = no pain; 10 = worst possible pain). | Evaluation will be done within three hours before image acquisition (SPECT).
DN4 scale | Evaluation will be done within three hours before image acquisition (SPECT).
Brief Inventory Pain | Evaluation will be done within three hours before image acquisition (SPECT).
Hospital Anxiety and Depression (HAD) scale | Evaluation will be done within three hours before image acquisition (SPECT).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brefel-Courbon, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

REFERENCES:
- [Result] Dellapina E, Pellaprat J, Adel D, Llido J, Harroch E, Martini JB, Kas A, Salabert AS, Ory-Magne F, Payoux P, Brefel-Courbon C. Dopaminergic denervation using [123I]-FPCIT and pain in Parkinson's disease: a correlation study. J Neural Transm (Vienna). 2019 Mar;126(3):279-287. doi: 10.1007/s00702-019-01974-5. Epub 2019 Jan 31. PMID 30706197